CLINICAL TRIAL: NCT03809767
Title: A Phase Ia/Ib, Open-Label, Multiple-Dose, Dose-Escalation and Expansion Study of the Anti-PD-1 Monoclonal Antibody CS1003 in Subjects With Advanced Solid Tumors or Lymphomas
Brief Title: A Study of CS1003 in Subjects With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1003-102
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CS1003 monoclonal antibody (Experimental)
  Interventions: Drug: CS1003 monoclonal antibody

INTERVENTIONS:
Drug: CS1003 monoclonal antibody — CS1003 will be administered intravenously every 3 weeks.

SUMMARY:
This is a phase Ia/Ib, open-label, multiple-dose, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of CS1003 in subjects with advanced solid tumors or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the informed consent.
2. Subjects must have histologically or cytologically confirmed advanced or metastatic solid tumor or unresectable lymphoma and have progressed, are intolerant to, refuse to accept or do not have access to standard therapy.
3. ECOG performance status of 0 or 1.
4. Subjects with evaluable but non-measurable lesion are eligible for Phase Ia. Subjects must have at least one measurable lesion per RECIST Version 1.1 to be eligible for Phase Ib.
5. Archived tumor tissue samples need to be collected, or subjects consent to undergo pre-treatment biopsy if archived sample is not available.
6. Life expectancy ≥ 3 months.
7. Subject must have adequate organ function.
8. Use of effective contraception (males and females).

Exclusion Criteria:

1. Subjects with known symptomatic or untreated brain metastasis or other CNS metastasis.
2. Subjects with active autoimmune diseases or history of autoimmune diseases.
3. Subjects who have to receive glucocorticoids (prednisone at > 10 mg/day or equivalent) or other immunosuppression within 14 days prior to the first dose of CS1003.
4. Subjects with other malignant tumor(s) in the past 2 years are not eligible for Phase Ib
5. Subjects who have received any immune checkpoint treatment, including PD-1, PD-L1, etc.
6. History of HIV infection.
7. Subjects with active Hepatitis B and C infection requiring therapy.
8. Subjects with active infection of tuberculosis.
9. History of organ transplantation.
10. Unresolved toxicities from prior anti-cancer therapy.
11. History of uncontrolled allergic asthma and serious hypersensitive reaction to monoclonal antibodies.
12. Subjects with major cardiovascular diseases.
13. History of alcoholism or drugs abuse.
14. Any condition that, in the opinion of the investigator or sponsor, would jeopardize compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | from the day of first dose to 90 days after last dose of CS1003

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Beijing Cancer Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Yunnan Cancer Hospital, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai pulmonary hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou

REFERENCES:
- [Derived] Gong J, Guo Y, Zhang Y, Ba Y, Chen T, Li W, Zhou C, Wang M, Yang H, Zhou Y, Cai Q, Wang Z, Huang G, Zhang W, Su R, Cai Z, Yue Z, Dou J, Li P, Wu R, Tse AN, Shen L. A Phase 1a/1b Dose Escalation/Expansion Study of the Anti-PD-1 Monoclonal Antibody Nofazinlimab in Chinese Patients with Solid Tumors or Lymphoma. Target Oncol. 2024 Sep;19(5):723-733. doi: 10.1007/s11523-024-01091-8. Epub 2024 Sep 4. PMID 39231855
- [Derived] Gao Y, Hu S, Li R, Jin S, Liu F, Liu X, Li Y, Yan Y, Liu W, Gong J, Yang S, Tu P, Shen L, Bai F, Wang Y. Hyperprogression of cutaneous T cell lymphoma after anti-PD-1 treatment. JCI Insight. 2023 Feb 22;8(4):e164793. doi: 10.1172/jci.insight.164793. PMID 36649072